CLINICAL TRIAL: NCT07124572
Title: Construction and Application of Precise Diagnosis and Treatment System for Thyroid-associated Ophthalmopathy
Status: Recruiting | Type: Observational
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-0592
Record Dates: First submitted 2025-08-06; First posted 2025-08-15 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-07

CONDITIONS: Thyroid Associated Ophthalmopathy
MeSH Terms: conditions — Graves Ophthalmopathy | interventions — X-Rays

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Participants without Thyroid-associated ophthalmopathy: Participants without thyroid-associated ophthalmopathy based on Bartley criteria.
  Interventions: Other: Imaging and ocular examinations
- Patients with Thyroid-associated ophthalmopathy: Patients diagnosed as thyroid-associated ophthalmopathy based on Bartley criteria.
  Interventions: Other: Imaging and ocular examinations

INTERVENTIONS:
Other: Imaging and ocular examinations — 2D and 3D Facial photography, blinking videos, orbital CT and MRI images, fundus images and images of nine gaze positions are taken.
  Clinical information is recorded. Quality of life is assessed. Ocular examinations, such as visual acuity, levator function, exophthalmos measurement, strabismus test, visual field examination, axial length measurement, OCT, OCTA are made.

SUMMARY:
This study aims to develop the deep learning-based system that integrates multimodal information to automatically diagnose, stage, and grade thyroid-associated ophthalmopathy (TAO), assist in treatment decision-making, and predict patient prognosis, thereby providing novel tools to support clinical management.

ELIGIBILITY:
Inclusion Criteria:

* normal participants without eyelid disorders (control group)
* patients with thyroid-associated ophthalmopathy (TAO group)
* cooperative participants

Exclusion Criteria:

* participants with pupil or cornea disorders
* participants with history of eye injury

Ages: 7 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: 500 patients with thyroid-associated ophthalomopahty 500 patients without thyroid-associated ophthalomopahty
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2030-10-01 (Estimated); Study Completion 2031-10-01 (Estimated)

PRIMARY OUTCOMES:
eye morphological parameters | through study completion, average of 5 years
  Margin reflex distances(mm)
Blinking feature of patients with thyroid-associated ophthalmopathy | through study completion, average of 5 years
  Blinking frequency
Ocular movement measurement | through study completion, average of 5 years
  Ocular movement ability in nine gaze positions
Automatic orbital structures segmentation and measurement using deep learning methods | through study completion, average of 5 years
  Automatic segmentation and measurement of orbital structures,such as eyeball, extraocular muscle, orbital fat, bony orbital region, optic nerves, etc
Automatic diagnosis, grading, staging and prediction of patients with thyroid-associated ophthalmopathy | through study completion, average of 5 years
  Patients with thyroid-associated ophthalmopathy(TAO) are classified as TAO or non-TAO. Grading is classified as mild, moderate, severe and sight-threatening. Staging is classified as active and stable.
three-dimensional eye parameters | through study completion, average of 5 years
  eyelid volume

CONTACTS AND LOCATIONS:
Locations (1):
- Juan Ye, Hangzhou, Zhejiang, China